CLINICAL TRIAL: NCT05749094
Title: The Sonographic Assessment of the Optic Nerve Sheath in Giant Cell Arteritis
Brief Title: Optic Nerve Sheath Ultrasound in Giant Cell Arteritis
Acronym: SONIC-GCA
Status: Recruiting | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Ciusss de L'Est de l'Île de Montréal (Other); Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke (Other); Mount Sinai Hospital, Canada (Other); St. Joseph's Health Care London (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jean-Paul Makhzoum, Director - Vasculitis Research Program, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 20201890
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Giant Cell Arteritis; Anterior Ischemic Optic Neuropathy; Optic Neuropathy, Ischemic
MeSH Terms: conditions — Giant Cell Arteritis; Optic Neuropathy, Ischemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA group: Ascertainment of GCA will occur 6 months after study inclusion and will require all the following features: 1) initial symptoms and clinical evolution consistent with GCA; 2) at least one positive diagnostic test for GCA, including ultrasound of temporal arteries, temporal artery biopsy, cranial MRI or cranial PET; and 3) satisfies the 2022 ACR-EULAR classification criteria for GCA.
  Study visits :
  Baseline - Month 3, 6, 12, 18 and 24 + relapse visit (if applicable)
  Interventions: Diagnostic Test: Optic nerve sheath ultrasound; Diagnostic Test: Standardized GCA assessment
- Non-GCA group: Participants who do not meet the composite clinical test validation for GCA (above).
  Study visits : Baseline and Month 6 (phone follow-up)
  Interventions: Diagnostic Test: Optic nerve sheath ultrasound; Diagnostic Test: Standardized GCA assessment

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath ultrasound — The patients are examined in a supine relaxed position. The probe is gently placed on the closed eyelid with a standard ultrasound gel and adjusted to a suitable angle to display the optic nerve entry into the eyeball. Measurements are done 3mm distal to the posterior aspect of the ocular globe. Ultrasosonographic 14L5 probe is used with a safe thermal index, mechanical index and intensity limit. All patients will also undergo a bedside fundoscopic examination. Official ophthalmology consultation will be requested in patients with visual symptoms or abnormal fundoscopy.
Diagnostic Test: Standardized GCA assessment — Clinical assesment, blood test review, temporal/axillary artery ultrasound

SUMMARY:
The Sonographic Assessment of the Optic Nerve Sheath in Giant Cell Arteritis (SONIC-GCA) study will evaluate the performance of the optic nerve sheath diameter (ONSD), measured via ultrasound, to diagnose and monitor GCA. SONIC-GCA builds upon our previous pilot studies and will answer the following questions:

1. What is the performance of ONSD to identify patients with new-onset, active GCA?
2. Is ONSD useful for monitoring GCA relapses during follow-up?
3. What is the intra- and interobserver reliability of ONSD measurements?
4. Does ONSD differ between patients with and without GCA-related retinal findings?

DETAILED DESCRIPTION:
SONIC-GCA is a prospective cohort and validation study conducted in centers of the Canadian Vasculitis Research Network (CanVasc).

ELIGIBILITY:
Our population of interest is patients referred from any settings for suspected, new-onset GCA.

Inclusion criteria:

To be included in SONIC-GCA, participants must meet all the following criteria:

1. Age > 50 years.
2. Referral to a GCA clinic for suspected, new-onset GCA.
3. Ability to understand and willingness to sign an informed consent form.
4. Willingness to comply with study visits and procedures.

Exclusion criteria:

An individual who meets any of these criteria will be excluded from SONIC-GCA:

1. Referral for a suspected GCA relapse.
2. Current use of systemic glucocorticoids, with the following duration at the baseline visit: ≥ 14 consecutive days of oral glucocorticoids in the previous 30 days, or ≥ 7 consecutive days of oral glucocorticoids if intravenous glucocorticoids were administered in the previous 30 days.
3. Current use of any conventional or biologic immunosuppressive therapy.
4. Known previous medical history of retinal diseases, optic nerve diseases, demyelinating diseases, normotensive hydrocephalus, intracranial tumors (benign or malignant), or any conditions associated with intracranial hypertension.
5. Any condition that impairs the ability to perform optic nerve sheath ultrasound or fundoscopy.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants referred for suspected new-onset GCA.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of ONSD to identify new-onset GCA | Baseline
  The primary outcome of SONIC-GCA is to determine the optimal ONSD cutoff for identifying GCA at the baseline visit and to assess its diagnostic performance, including sensitivity, specificity, positive and negative predictive values, and accuracy.
ONSD in patients with and without GCA | Baseline
  At baseline, ONSD measurements (in mm) of the left and right eyes of each participant will be recorded and used to calculate the mean ONSD for patients with and without GCA.

SECONDARY OUTCOMES:
ONSD changes over time | Up to 2 years
  The main secondary outcome will determine whether ONSD dynamically correlates with relapse risk over the follow-up period in patients with GCA, providing insight into its potential as a biomarker for disease monitoring.
The associations between ONSD changes and GCA relapses | Up to 2 years
  The association between ONSD changes and GCA relapses will be assessed during the follow-up period, in patients with GCA.
Evaluation of the performance of ONSD to detect a GCA relapse | Up to 2 years
  We will assess the diagnostic performance of the initial ONSD cutoff (from the primary objective) at each follow-up visit to differentiate between relapse and remission. This analysis will determine whether the established cutoff remains a reliable marker for monitoring disease status in GCA over time.

OTHER OUTCOMES:
Intra- and Inter- observer reliability | Baseline
  Intra- and interobserver reliability of ONSD measurements
Association between ONSD and Retinal Changes | Up to 2 years
  The association between ONSD and the presence/absence of GCA-related retinal findings on digital fundoscopy in patients with GCA.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Makhzoum, MD, Study Chair — Vasculitis Clinic, Hopital du Sacre-Coeur de Montreal, University of Montreal
Locations (6):
- Canada (6):
  - St-Joseph's Health Care London, London, Ontario
  - Sinai Health - Toronto, Toronto, Ontario
  - MUHC - McGill University, Montreal, Quebec
  - Vasculitis Clinic, Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CIUSSS de l'Est-de-l'ile de Montreal, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vasculitis Clinic - University of Montreal — http://vasculitemontreal.com